CLINICAL TRIAL: NCT01779752
Title: Functional Organisation of the Vestibular Cortical Pathways in Human: Transcranial Magnetic Stimulation (TMS) Approach
Brief Title: Vestibular Cortex and TMS
Acronym: CoVest
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C12-20; 2012-A00839-34 (Registry Identifier: IDRCB)
Record Dates: First submitted 2013-01-17; First posted 2013-01-30 (Estimated); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Cortical Organisation of Vestibular Integration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In human, the cerebral cortex forms a network of vestibular cortical areas which functional role remains unknown. In patients with localised cortical lesions the investigator has previously demonstrated that the parieto-temporal cortex could regulate the inertial component of the vestibulo-ocular (VOR) responses whereas more ventral regions including the temporo-occipital cortex would be associated with gain regulation of these VOR responses.

The investigator's main purpose is to investigate the modalities of vestibular integration in these posterior parieto-temporal et temporo-occipital cortical regions. Thus, by using repetitive ttranscranial magnetic stimulation (rTMS) the investigator will induce a transitory inhibition of one of these 2 cortical regions and register its effect on VOR responses. Based on theta burst stimulation (TBS) paradigm, the investigator will stimulate the region of interest by applying on the scalp repetitive burst (at 50 HZ) during 44sec. Then, during the consecutive cortical inhibition lasting for the 15 minutes poststimulation, the investigator will record the subject's VOR responses. The VOR gain will be calculated and the time constant and phase will provide an estimation of the inertial component of the VOR responses. The healthy subjects recruited on the basis of inclusion criteria during medical examination will be divided into two groups of 20 subjects each depending of their sites of stimulation, temporo-parietal or temporo-occipital. Each subject will perform three experimental sessions (of 1h in average each) separated by at least one week and corresponding to : (1) the right cortical stimulation, (2) the left stimulation and (3) the vertex stimulation serving as the control session.

The TMS paradigm is used in routine in hospital and research field and had very few negative consequences (mainly transitory and occasional headache).

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female healthy volunteers between 20 and 35 years old.
* Considered healthy subject after medical examination and MRI images analysis
* With social security affiliation
* After informed and voluntary consent to participate to the study (signed written consent)
* With normal ocular responses with a gain not less than 0.5 during preliminary VOR registration.

Exclusion Criteria:

* Persons under guardianship, curatorship or any other administrative or judicial deprivation of rights and freedom
* Persons with a medical history, or any acute or chronic disease which may affect the test results, or creating a risk to the subject in the protocol, in particular:

  * with personal or family history of seizure disorders
  * with previous or current psychiatric disease or schizotypal signs (RISC questionary)
  * with previous or current neurology or otology (audition or equilibrium) history
  * with visual corrected visual acuity inferior to 8/10
  * having taken hypnotics, psychotropic or other central nervous system depressants (opiates, barbiturates, antiepileptics, antidepressants, sedatives, antihistamines, anxiolytics, neuroleptics, clonidine and related) during the 8 months prior to experimentation
  * consuming more than 150 mg of caffeine per day (15 small cups of Italian coffee)
  * with a contra-indication for MRI: pacemaker or neural surgical clips ferromagnetic and metallic implants, intraocular foreign bodies, claustrophobia
  * pregnancy (diagnosed by a urine test)

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Subjects
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2013-01-20 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
changes in gain of vestibulo-ocular reflex (VOR) | Day 1, Day 7, Day 14, Day 21